CLINICAL TRIAL: NCT03946644
Title: Comparison of Two Different Safety Distances to Sapheno-femoral Junction for EndoVenous Laser Ablation Treatment of Great Saphenous Vein Incompetence: a Prospective Randomized Double-blind Study
Brief Title: Safety Distance for Endovenous Laser Ablation of the Great Saphenous Vein
Acronym: SDEVLA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stanislava Tzaneva, Principal Investigator, Clinical Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 62018
Record Dates: First submitted 2019-01-23; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Great Saphenous Vein Incompetence; Endovenous Laser Ablation
Keywords: Safety distance; Laser ablation; Great saphenous vein

STUDY DESIGN:
Intervention Model Description: At day 0 (day of EVLA), 7-14 days after inclusion of the patients, patients will be randomized with the online randomization program "Randomizer" (https://www.meduniwien.ac.at/randomizer/web/login.php).Patients will be randomized to one of the following two groups:
  * EVLA with keeping of security distance of 2cm to the SFJ
  * EVLA without keeping a distance tot he SFJ
Who Masked: Participant, Investigator
Masking Description: The blinding of the patients is facilitated by the same mode schedule and the same treatment performance for both allocations.
  The patients will not be informed of their treatment allocation. The clinical investigator who will prepare the follow-up investigations will not have information about treatment allocation too. The blinded investigator will not have access to the full documentation of the study and to randomizing data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVLA with keeping of security distance (Active Comparator): The EVLA will be performed with the 1470nm diode laser and a radial fibre (Leonardo® - 1470 nm/15W, Biolitec). The exact position of the catheter tip will be fixed under ultrasound guidance 2 cm below the SFJ.
  Interventions: Device: EVLA with keeping of securuty distance
- EVLA without keeping a distance (Experimental): The EVLA will be performed with the 1470nm diode laser and a radial fibre (Leonardo® - 1470 nm/15W, Biolitec). The exact position of the catheter tip will be fixed under ultrasound guidance without keeping a distance to the SFJ.
  Interventions: Device: EVLA without keeping a distance

INTERVENTIONS:
Device: EVLA with keeping of securuty distance — The EVLA will be performed with the 1470nm diode laser and a radial fibre (Leonardo® - 1470 nm/15W, Biolitec). The exact position of the catheter tip will be fixed under ultrasound guidance 2 cm below the SFJ.
  Arms: EVLA with keeping of security distance
Device: EVLA without keeping a distance — The EVLA will be performed with the 1470nm diode laser and a radial fibre (Leonardo® - 1470 nm/15W, Biolitec). The exact position of the catheter tip will be fixed under ultrasound guidance without keeping a distance to the SFJ.
  Arms: EVLA without keeping a distance

SUMMARY:
Chronic venous disease is one of the most common diseases in the western world and worldwide with a prevalence of 83,6%. It is a chronic progressive disease, which causes a significant burden on health systems, treatment and care of these patients. Recurrence of varicose veins after successful treatment remains a problem and has been reported in up to 30% of patients after endovenous laser ablation (EVLA), which is the recommended treatment of choice for incompetence of the truncal veins. The aim of this project is to investigate a variation of the EVLA, which has the potential to reduce the recurrence rate in the long-term. If this assumption is true, the investigators expect reduction of costs in the health system and improved quality of life for individual patients.The primary objective of the project is the evaluation of long-term anatomical effectiveness of EVLA treatment with and without keeping a distance to sapheno-femoral junction (SFJ), defined as complete obliteration of the great saphenous vein (GSV) or absence of an open saphenous stump at the SFJ after 3 years. Secondary objectives are:

1. . Evaluation of the effectiveness of EVLA treatment with and without keeping a distance to SFJ, measured as duplex sonographic reflux (≥ 0,5 sec) in the GSV or any other axial vein at the SFJ after 1 year and 3 years.
2. . Evaluation of the anatomical effectiveness of EVLA treatment with and without keeping a distance to SFJ, measured as the length of the open saphenous stump (in centimeters) after 1 year and 3 years.
3. . Assessment of quality of life 3 months, 1 year and 3 years after EVLA.
4. . Evaluation of the clinical efficacy and tolerability measured as a clinical score at 3 months, 1 year and 3 years after EVLA.
5. . Safety assessment measured as the number of thromboembolic events 1 week and 3 months after EVLA.This project is planned as a prospective randomized parallel group double-blind study.

For the assessment of efficacy and safety parameters, clinical examinations and duplex sonographic examinations will be performed 3 months, 1 year and 3 years after the intervention.

For the assessment of tolerability endpoints, clinical scores and quality of life score will be performed 3 months, 1 year and 3 years after EVLA. Clinical scores include Clinical, Etiologic, Anatomical, and Pathophysiological Classification (CEAP) and Venous Clinical Severity Scoring (VCSS) and for evaluation of quality of life Aberdeen Varicose Veins Questionnaire (AVVQ) will be used.

DETAILED DESCRIPTION:
Introduction and background information Chronic venous disease is one of the most common diseases in the western world and worldwide with a prevalence of 83,6%. It is a chronic progressive disease, which causes a significant burden on health systems, treatment and care of these patients.

There are different methods for treatment of insufficiency of the GSV, which have good evidence: open surgery and minimally invasive techniques including ultrasound-guided foam sclerotherapy (UGFS), radiofrequency ablation (RFA) and endovenous laser ablation (EVLA). UGFS and thermal ablation techniques such as EVLA have become widely used alternatives to surgery for the treatment of venous reflux. The safety and efficacy of EVLA has been demonstrated in several studies. According to guidelines of the European Venous Forum (EVF), the International Union of Angiology (IUA) and the European Society for Vascular Surgery (ESVS) the treatment of GSV reflux with EVLA is recommended in preference to surgery, Grade of Recommendation 1A.

Rationale of the project Recurrence of varicose veins after successful treatment remains a problem and has been reported in up to 30% of patients after EVLA. Treatment with EVLA aims at complete obliteration of the vein in the treated area. According to the literature a safety distance of 1-2 cm from the sapheno-femoral junction (SFJ) is obligatory in all patients undergoing EVLA of the GSV. In earlier trials laser systems equipped with a bare fibre were used, which emit shorter wavelength of 810 nm antegrade with an absorption maximum in the range of haemoglobin. A new generation of laser devices with a wavelength of 1470 nm has been introduced in recent years. The absorption coefficient of water at 1470 nm is significantly higher than in the wavelength range of 810 - 1064 nm, which results in a much better control of the laser energy applied. The patented radial (360°) fibre ensures radial delivery of energy inducing homogenous photothermal destruction of the vein wall. By avoiding perforation of the vein wall and associated thermal irritation of the surrounding tissue, post-operative pain is minimized, as are ecchymosis and other side effects noticed with the previously used bare fibres.

In prospective studies it has been demonstrated that EVLA of the GSV using radial fibres has fewer side effects compared to EVLA of the GSV using bare fibre. It is not known whether the use of radial fibres results in a complete vascular closure of GSV up to the SFJ, and whether a remaining non-occluded vessel stump could be a cause of recurrence. Applying EVLA without keeping a distance of 1-2 cm to the SFJ is used with increasing frequency by many specialists, but there is no controlled data about this topic.

At our department the investigators use a 1470 nm laser with radial fibres without keeping a distance to SFJ and have no complications observed so far.

The aim of this project is to compare the efficacy and safety parameters when two different distances from the SFJ during EVLA of the GSV are kept. Our scientific hypothesis is that EVLA of the GSV with placing the catheter tip at the SFJ without keeping a distance to the SFJ leads to better anatomical results (complete obliteration of the GSV) after three years compared to EVLA with keeping a distance of 2 cm from the SFJ. If this hypothesis is true, a reduction in the incidence of recurrent varicose veins after EVLA of the GSV would be expected when placing the catheter tip without keeping a distance to the SFJ. This risk reduction would have a positive impact on patient quality of life and on the consumption of resources in the health system.

Objectives of the project (hypothesis)

Primary objective:

The primary objective of the study is the complete anatomical obliteration rate of the ablated GSV or absence of an open saphenous stump 3 years after EVLA in both groups.

Null hypothesis: EVLA without keeping a distance to the SFJ does not result in an equal obliteration rate of the GSV or absence of an open saphenous stump 3 years after surgery compared to EVLA with maintaining a distance to the SFJ of 2 cm.

Alternative hypothesis: EVLA without keeping a distance to the SFJ results in an equal obliteration rate of the GSV or absence of an open saphenous stump 3 years after surgery compared to EVLA with maintaining a distance from the SFJ of 2 cm.

Secondary objectives are:

Complete obliteration rate of the GSV or absence of an open saphenous stump 1 year after EVLA in both groups Duplex sonographic reflux (≥0,5 sec) in the GSV or any other axial vein at the SFJ 1 and 3 years after EVLA Length of the open saphenous stump (in centimetres) 1 year and 3 years after EVLA Clinical efficacy and tolerability measured as a clinical score 3 months, 1 year and 3 years after EVLA Overall quality of life 3 months, 1 year and 3 years after EVLA Overall safety measured as the number of thromboembolic events 1 week and 3 months after EVLA Design of the clinical investigation Prospective, randomized, parallel group, double blind study Population Subject population: Patients with incompetence of the GSV that have been referred to the phlebologic-angiological unit of the Division of General Dermatology and Dermato-Oncology, Medical University of Vienna Methodology Measurements and analysis Eligibility and Enrolment Study team will ensure that patients meet the criteria for study enrolment. Patients must consent to screening for eligibility. Enrolment will occur after eligibility is established and informed consent is provided.

Screening In all patients, past history will be collected including drug history. There will be a physical examination including height- and body weight measurements. All patients will be examined clinically and by duplex sonography prior to EVLA. Inclusion and exclusion criteria will be checked.

Clinical examination Clinical, etiologic, anatomic, pathophysiology (CEAP) classification will be performed at screening and by a blinded investigator at the baseline examination, as well as during the follow-up period at 3 months, 1 and 3 years. The Venous Clinical Severity Score (VCSS) will be also determined at screening and by a blinded investigator at baseline, 3 months, 1 year and 3 years post procedure.

A blinded investigator will clinically examine all patients 1 week postoperatively, 3 months, 1 year and 3 years after EVLA.

Quality of life All patients, who are eligible to enter the study, will fill in a questionnaire for quality of life.

The quality of life will be determined by means of Aberdeen Varicose Vein Questionnaire (AVVQ) at baseline and 3 months, 1 year and 3 years after EVLA. The questions will be answered by the patient and documented by a blinded investigator at baseline and after 3 months, 1 year and 3 years; see Table 1.

Duplex sonographic examination Duplex scanning investigation (LOGIQ® 7 General Electric Austria GmbH) will be performed at screening to establish the diagnosis of incompetence of the GSV and to check the inclusion and exclusion criteria for eligibility. Follow-up investigation will be performed 1 week postoperatively, 3 months, 1 year and 3 years after EVLA. During the trial a blinded investigator without knowledge of the patient group will perform the duplex ultrasound examination. If a diagnosis of EHIT or venous thromboembolic events (VTE) is made, weekly duplex sonographic controls will be performed until resolving of EHIT.

EVLA will be performed in local tumescent anaesthesia or general anaesthesia depending on the patient's preference and clinical findings. Treatment will be performed on an inpatient basis.

This procedure will be performed with the patient and all people in the room wearing protective eye goggles to guard against unplanned exposure to the laser.

The EVLA will be performed with the 1470nm diode laser and a radial fibre (Leonardo® - 1470 nm/15W, Biolitec). The GSV will be punctured with an 18-gauge needle under sonographic guidance and the laser fibre will be introduced by Seldinger technique at the distal point of insufficiency, possibly no deeper than the proximal tibia. The laser catheter will be advanced forward to the SFJ. The exact position of the catheter tip will be fixed under ultrasound guidance depending on randomization, either without keeping a distance to the SFJ or 2 cm below the SFJ. Thereafter, the saphenous vein will be overmolded with tumescence (in patients with tumescent anaesthesia) or saline (in patients with general anaesthesia) also under ultrasound guidance. The laser energy will be administered under continuous pull back of the catheter in a total dose of 80J /cm2 and 10W/cm2. EVLA will be applied only for the GSV. In the same session insufficient side branches will be removed by phlebectomy.

Both the patient and the investigator will be blinded with respect to the treatment group.

After EVLA compression stockings class 2 (25-35 mm Hg) will be applied for a week during day and night. Patients will be advised to wear tight length compression stockings class 2 for another 3 weeks daytime if additional phlebectomias have been performed. The patient should move around a lot and drink enough, at least 2 litres per day. Heat procedures such as hot baths, thermal baths, sauna, solarium, and direct exposure to sunlight should be avoided for the duration of 4-6 weeks after the procedure. Short shower with lukewarm water is allowed.

Analgetics and NSAIDs upon need are postoperatively allowed. In patients at thrombotic risk Low Molecular Weight Heparin (LMWH) in prophylactic dose will be administered for at least 1 week and for a maximum of 6 weeks after EVLA depending on individual risk. The following patients are classified as risk patients: patients with chronic inflammatory diseases, patients with cancer, patients with previous thromboembolic events, thrombophilia patients, patients with obesity, patients on estrogen-containing oral contraceptives or hormone replacement therapy and immobilization postoperatively for different reasons.

Follow-up Follow-up investigations will be carried out 1 week, 3 months, 1 year and 3 years after EVLA. If a diagnosis of EHIT or VTE is made, weekly duplex sonographic controls will be performed until resolving of EHIT.

All patients will undergo physical and duplex sonographic examination 1 week postoperatively. All adverse events and complaints of the patients will be documented in the CRF at every follow-up visit. At 3 months follow up every patient will be examined clinically with determination of CEAP and VCSS and duplex sonographic as described above, methodology, duplex sonographic examination. The Quality of life will be determined by means AVVQ and clinical photographs will be taken. These investigations will be repeated 1 year and 3 years after EVLA.

ELIGIBILITY:
Inclusion Criteria:

1. . Age ≥ 18 years
2. . Duplex sonographic reflux in GSV ≥ 0,5 seconds
3. . Straight run of the GSV in the thigh

Exclusion Criteria:

1. . Acute thromboembolic events
2. . Active cancer
3. . Postthrombotic syndrome from obstruction type
4. . Severe peripheral arterial occlusive disease (PAOD, ankle brachial index (ABI) ≤ 0.5)
5. . Pregnancy and breast feeding
6. . Incompetence of the anterior accessory great saphenous vein (AAGSV)
7. . Intolerance for compression stockings
8. . Contraindications for local anesthesia or general anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2018-09-26 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of Complete obliteration of the GSV or absence of an open saphenous stump at the SFJ 3 years after EVLA | 3 years
  Number of complete obliteration of the GSV or absence of an open saphenous stump will be assessed by duplex-sonographic investigation

SECONDARY OUTCOMES:
Number of GSV with Duplex sonographic reflux (≥ 0,5 sec) or any other axial vein at the SFJ | 1 year and 3 years
  Number of GSV or any other axial veins with duplex sonographic reflux measured by duplex-sonographic investigation. Reflux is defined as equal or longer than 0,5 sek
Length of the open saphenous stump (in centimeters) | 1 year and 3 years
  The length of the open saphenous stump will be measured by duplex-sonographic investigation
Satisfaction assessed by the QOL | 3 months, 1 year, 3 years
  Patients' satisfaction will be assessed by using standardized quality of life questionnaire named Aberdeen varicose vein questionnaire. The questionnaire consist of 13 questions relating to all aspects of the problem of varicose veins, is scored from zero to 100, were zero represents a patient with no evidence of varicose veins and 100 represents the most severe problems associated with varicose veins.
points of Clinical score | 3 months, 1 year, 3 years
  Evaluation of the clinical efficacy and tolerability measured as a clinical score by means of Venous Clinical Severity Score (VCSS) scale, maximal score of 30 points. The VCSS includes 9 hallmarks of venous disease, each scores on a severity scale from 0 to 3.
Incidence of treatment-emergent adverse events assessed as Number of thromboembolic events | 1 week, 3 months
  Number of thromboembolic events will be assessed by duplex sonographic examination.

CONTACTS AND LOCATIONS:
Overall Officials: Stanislava Tzaneva, MD, Principal Investigator — University Clinic of Dermatology
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No